CLINICAL TRIAL: NCT04208672
Title: Validation of a Handy Sleep Monitoring Device: UMindSleep in Patients With Obstructive Sleep Apnea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Zhang Jihui, Assistant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CREC2018.501
Record Dates: First submitted 2019-09-03; First posted 2019-12-23 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Validation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient attending for PSG in Sleep Assessment Unit (Experimental): Subjects referred to the SAU will be invited to participate into this study
  Interventions: Device: UMindSleep

INTERVENTIONS:
Device: UMindSleep — CPAP titration will be provided for Obstructive Sleep Apneas Syndrome.

SUMMARY:
This is a validation study recruiting subjects with and without obstructive sleep apnea. All subjects will undergo a nocturnal standard polysomnography and UMindSleep assessment. Sleep parameters, such as sleep stages and apnea UMindSleep software. Correlation in each parameter between PSG and events in polysomnography (PSG) will be scored according to the AASM criteria while the sleep parameters will be automatically scored by the UMindSleep will be analyzed to determine the magnitude of agreement between UMindSleep and PSG.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a common sleep disorder in the general population with a prevalence ranging from 4-30%. OSA has been shown to be a significant risk factor of many cardiovascular diseases and mental disorders. However, OSA is a neglected problem in the general population. In addition, there is a significant unmet need for the treatment of OSA. One of the major reason for the under-diagnosis and under-treatment of OSA in the general population is a lack of reliable screening tool in detecting OSA. In this regard, several devices, such as ApneaLink, have been developed for the screening of OSA. However, as this kind of device only employs time in bed rather than actual sleep time to calculate the apnea index or desaturation index, they tend to underestimate the severity of sleep apnea. In this regard, it is timely need to develop and validate new device that can integrate the actual sleep time and apnea or desaturation events for the precise calculation of sleep apnea index or desaturation index.

The UMindSleep is a handy and wearable device to acquire EEG, heart rate, saturation, snoring and temperature. The signal will be uploaded to a smartphone through Bluetooth. By integrating these signals, the system can automatically analyze several key parameters by the algorithms, such as sleep stages and desaturation events.

ELIGIBILITY:
Inclusion Criteria:

* complain of habitual snoring;
* AHI as measured by standard PSG > 5/hour

Exclusion Criteria:

* Aged 17 years old or below
* patients with narcolepsy and REM sleep behavior disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-01-16 (Estimated); Primary Completion 2020-03-15 (Estimated); Study Completion 2020-09-15 (Estimated)

PRIMARY OUTCOMES:
sleep apnea | 6 months
  The correlation of Sleep staging and Apnea-hyponea index measured by PSG and UMindSleep will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of psychiatry, Faculty of Medicine, The Chinese University of Hong Kong, Hong Kong, Hong Kong